CLINICAL TRIAL: NCT01908933
Title: Study of the AeriSeal System Treatment in Patients With Advanced Non-Upper Lobe Predominant Heterogeneous Emphysema
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-C13-001PLV
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Advanced Emphysema; Heterogeneous Lower Lobe Predominant Emphysema; Heterogeneous Upper and Lower Lobe Predominant
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AeriSeal Emphysematous Lung Sealant Syst (Experimental): This is a prospective, open label, single-arm, multicenter, investigational study. Patients will receive either unilateral or bilateral AeriSeal System therapy as appropriate utilizing 20 mL/subsegment dosing at 2 to 4 subsegments.
  Interventions: Device: AeriSeal Emphysematous Lung Sealant Syst

INTERVENTIONS:
Device: AeriSeal Emphysematous Lung Sealant Syst — This is a prospective, open label, single-arm, multicenter, investigational study. Patients will receive either unilateral or bilateral AeriSeal System therapy as appropriate utilizing 20 mL/subsegment dosing at 2 to 4 subsegments.

SUMMARY:
The purpose of this study is to prospectively evaluate the safety and efficacy of the AeriSeal System in patients with advanced Non-Upper Lobe Predominant Heterogeneous Emphysema.

DETAILED DESCRIPTION:
This is a prospective single arm study to evaluate the safety and efficacy of the AeriSeal System in patients with advanced Non-Upper Lobe Predominant Heterogeneous Emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and to participate in the study
* Age > or = 40 years at the time of the screening
* Advanced lower or lower and upper lobe predominant heterogeneous emphysema by CT scan
* Minimum of 2 subsegments appropriate for treatment
* MRCD questionnaire score of 2 or greater at screening
* Failure of medical therapy to provide relief of symptoms
* Spirometry 15 minutes after administration of bronchodilator (BOTH):

  * FEV1 < 50 % predicted.
  * FEV1/FVC ratio <70 %
* Lung volumes by plethysmography (BOTH):

  * Total Lung Capacity (TLC) > 100 % predicted
  * Residual Volume (RV) > 150 % predicted
* Diffusing Capacity of Carbon Monoxide(DLco) > = 20 and < = 60 percent predicted
* Oxygen saturation (SpO2) > 90 % on < or = 4 L/min supplemental O2, at rest
* Six-Minute Walk Test distance > or = 150 m
* Abstinence from smoking for at least 16 weeks prior to screening

Exclusion Criteria:

* Prior lung volume reduction surgery, prior lobectomy or pneumonectomy, or prior lung transplantation
* Requirement for ventilator support (invasive or non-invasive)
* Three (3) or more COPD exacerbations requiring hospitalization within 1 year of Screening visit or a COPD exacerbation requiring hospitalization within 8 weeks of Screening visit
* Pulmonary hypertension, defined as:

  * Echocardiogram with estimated peak systolic pressure > 45 mmHg in the presence of tricuspid valve regurgitation stated in the echocardiogram report
  * If the echocardiogram shows peak systolic pressure > 45 mmHg, right heart catheterization is required to rule out pulmonary hypertension, defined as peak systolic pressure > 45 mmHg or mean pressure > 35 mmHg
* Clinically significant asthma (reversible airway obstruction) or bronchiectasis
* CT scan: Presence of the following radiologic abnormalities:

  * Pulmonary nodule on CT scan greater that 1.0 cm in diameter (Does not apply if present for 2 years or more without increase in size or if proven benign by biopsy/PET)
  * Radiologic picture consistent with active pulmonary infection, e.g., unexplained parenchymal infiltrate
  * Significant interstitial lung disease
  * Significant pleural disease
  * Giant bullous disease (a predominant bulla > 10 cm in all dimensions >1 / 3 of the hemithorax)
* Use of systemic steroids > 20 mg/day or equivalent, immunosuppressive agents, heparins, oral anticoagulants (e.g., warfarin, dicumarol; note: antiplatelet drugs including aspirin and clopidogrel are permitted)
* Allergy or sensitivity to medications required to safely undergo AeriSeal System treatment
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to the screening visit
* Body mass index < 15 kg/m2 or > 35 kg/m2
* Female patient pregnant or breast-feeding or planning to be pregnant in the next year
* Significant comorbidity that carries prohibitive risks or is associated with less than 2-year expected survival, including any of the following:

  * HIV/AIDS
  * Active malignancy
  * Stroke or Transient Ischemia Attack (TIA) within 12 months of screening
  * Myocardial infarction within 12 months of screening
  * Congestive heart failure within 12 months of screening defined at clinical evidence of right or left hear failure or left ventricular ejection fraction < 45 % on echocardiogram
* Any condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the patient such as alcoholism, high risk for drug abuse or noncompliance in returning for follow-up visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Volume change by CT | 28 - 30 weeks
  Group mean normalized change from baseline in the volume of the treated lung lobes measured by quantitative CT at 24 weeks post-treatment (defined as the sum of volume change in all treated lobes/number of treatments).

SECONDARY OUTCOMES:
Fraction of patients showing clinically significant improvements from baseline in one or more of the following outcomes at 24 weeks post treatment: Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), Medical Research Council Dyspnea | 28 - 30 weeks
  Group mean change in baseline to week 24 in:Forced Expiratory Volume in 1 second (FEV1),Forced Vital Capacity (FVC),Medical Research Council Dyspnea (MRCD), 6 Six-Minute Walk Test (6MWT), Saint George Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, Prof. Dr med, Principal Investigator — Thoraxklinik am Uniklinikum Heidelberg; Wolfgang Gesierich, Dr med, Principal Investigator — Asklepios Fachkliniken Muenchen - Gauting; Manfred Wagner, Dr med, Principal Investigator — Klinikum Nuernberg Nord; Mordechai Kramer, Prof, Principal Investigator — Rabin Medical Center; Martin Hetzel, Dr med, Principal Investigator — Krankenhaus vom Roten Kreuz - Stuttgart